CLINICAL TRIAL: NCT00607932
Title: Effects of Bassica or Indole-3-Carbinol on Prostatectomy Patients With PSA Recurrence
Brief Title: Brassica Vegetables or Indole-3-Carbinol in Treating Patients With PSA Recurrence After Surgery for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jay Fowke, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000581410; VU-VICC-URO-0369; VU-VICC-041001
Record Dates: First submitted 2008-02-01; First posted 2008-02-06 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — indole-3-carbinol; Counseling; Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brassica Vegetables Diet Intervention (Experimental)
  Interventions: Behavioral: behavioral dietary intervention; Dietary Supplement: Brassica vegetable; Drug: indole-3-carbinol; Other: counseling intervention; Other: medical chart review; Other: questionnaire administration; Procedure: adjuvant therapy
- Pill (Experimental)
  Interventions: Drug: indole-3-carbinol; Other: counseling intervention; Other: medical chart review; Other: questionnaire administration; Procedure: adjuvant therapy

INTERVENTIONS:
Behavioral: behavioral dietary intervention
  Arms: Brassica Vegetables Diet Intervention
Dietary Supplement: Brassica vegetable
  Arms: Brassica Vegetables Diet Intervention
Drug: indole-3-carbinol — follow up at 2,4,6 months post baseline.
  Other Names: I3C
Other: counseling intervention — 2, 4, 6 months post baseline
Other: medical chart review — 2,4,6 months post baseline
Other: questionnaire administration
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Eating a diet high in vegetables may lower the risk of some types of cancer. Brassica vegetables (such as cabbages, kale, broccoli, Brussels sprouts, and cauliflower) and indole-3-carbinol (a substance found in cruciferous vegetables) may help lower the risk of prostate cancer recurrence.

PURPOSE: This randomized clinical trial is studying the side effects and how well Brassica vegetables work compared with indole-3-carbinol in treating patients with PSA recurrence after surgery for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of Brassica vegetable intake and indole-3-carbinol supplement use in patients with prostate cancer with prostate-specific antigen (PSA) recurrence after prostatectomy.
* Identify adverse events in these patients.
* Quantify the effects of each intervention on PSA in these patients.

OUTLINE: Patients are stratified by pretreatment prostat-specific antigen (PSA) growth rate (low [0.00-0.15] vs medium [0.16-0.30] vs high [> 0.30]). They are randomized to 1 of 3 treatment arms, and randomization status to arms II and III is double-blinded.

* Arm I (Brassica vegetables): Patients consume Brassica vegetables at least 2 servings (½ cup/serving) daily for 6 months. Patients meet one-on-one with the study dietician, and are instructed on the potential health benefits of Brassica vegetables and purchase and preparation of the vegetables. Patients undergo telephone counseling periodically in months 1-5, to monitor their progress and identify barriers to adherence and to develop solutions to overcome these barriers.
* Arm II (Placebo): Patients receive oral placebo once daily for 6 months.
* Arm III (Indole-3-carbinol supplement): Patients receive oral indole-3-carbinol supplement (capsules) once daily for 6 months.

Blood and urine samples (for urinary isothiocyanate levels) are collected at baseline and at 2, 4, and 6 months. Patients complete questionnaires assessing demographics, family cancer history, and health history and measuring changes in medications, lifestyle, adverse events, and health. Medical records are reviewed for prostate cancer-related information, surgical dates, dose and type of radiation, and PSA history.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer with PSA recurrence after prostatectomy

  * PSA recurrence is defined as two consecutively rising PSA tests ≥ 8 weeks since the post-surgical nadir, with a minimal interval of 2 weeks between tests and at least 1 PSA test > 0.4 ng/mL

Exclusion Criteria:

* Life expectancy ≥ 9 months
* No predictors of poor adherence (e.g., erratic life-style, mental incompetence)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other concurrent Brassica vegetable consumption > 1 serving/day
* No other concurrent indole-3-carbinol supplements
* No endocrine or radiation treatment within past 4 weeks
* No other scheduled treatment during study intervention
* Concurrent prescription medications during the trial allowed

  * At least 2 weeks since prior and no concurrent vitamin or herbal supplement use

    * Patients refusing to stop non-study supplements will be asked to maintain constant use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of Brassica vegetable intake and indole-3-carbinol supplementation | will be measured at 2-Months, 4-Months, and 6-Months after Baseline start for the diet intervention
Adverse events | will be measured at 2-Months, 4-Months, and 6-Months after Baseline start for the diet intervention
Effects of intervention on prostate-specific antigen | Not noted

CONTACTS AND LOCATIONS:
Overall Officials: Jay H. Fowke, PhD, MPH, Study Chair — Vanderbilt-Ingram Cancer Center